CLINICAL TRIAL: NCT06642090
Title: Impact of Educational Programs on the Knowledge and Self-care of Patients Undergoing Hemodialysis in Morocco.
Brief Title: Educational Program for Patients Undergoing Hemodialysis.
Acronym: EDU-HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cadi Ayyad University (Other)
Responsible Party: Principal Investigator, MAZZI Loubna, Principal Investigator, Cadi Ayyad University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Semlalia-Hemodialysis-2024-001
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Hemodialysis; Self-care; End Stage Renal Disease
Keywords: Hemodialysis; Arteriovenous fistula self-care; Therapeutic adherence; Patient knowledge; Educational program
MeSH Terms: conditions — Kidney Failure, Chronic; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: This interventional study follows a randomized controlled trial (RCT) design, comparing the effectiveness of an educational intervention against standard care in patients undergoing hemodialysis. Participants will be randomly assigned to one of two groups: the intervention group, which will receive targeted educational sessions focused on chronic kidney disease management. The control group didn't receive any intervention.
  The educational program aims to enhance patient knowledge, improve self-management skills, and optimize clinical outcomes such as medication adherence and weight management. Assessments will be conducted at baseline and after the intervention to evaluate changes in knowledge, self-care behaviors, and clinical parameters.
  The study will be conducted in a public hemodialysis center in the Marrakech-Safi region, and aims to provide insights into the impact of educational interventions on patient outcomes in this population
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group: Standard Care in Hemodialysis (No Intervention): This arm of the study includes 34 patients undergoing hemodialysis who will notany intervention. Participants will continue to receive the usual care provided by the hemodialysis center. No educational sessions will be delivered in this group. Clinical outcomes, including health parameters, will be assessed in comparison to those in the intervention group after the study period.
- Intervention Group (Experimental): This intervention group includes 36 patients at a public hemodialysis center in the Marrakech-Safi region. this group will engage in an educational program designed to enhance their understanding of chronic kidney disease and promote self-care for venous access. The curriculum covers topics such as disease etiology, symptoms, hemodialysis principles, medication roles, and dietary recommendations. The ultimate objective is to improve treatment adherence and optimize the management of dry weight and interdialytic weight, surpassing the standard care received by the control group.
  Interventions: Behavioral: Educational intervention for patients undergoing hemodialysis in Morocco

INTERVENTIONS:
Behavioral: Educational intervention for patients undergoing hemodialysis in Morocco — This is the first educational intervention in Morocco to improve the knowledge, self-care, and biological characteristics of patients undergoing hemodialysis.
  Arms: Intervention Group

SUMMARY:
This study aims to evaluate the impact of an educational intervention on improving knowledge, self-care practices, and treatment adherence among hemodialysis patients at the Youssoufia Hemodialysis Center, located in the Marrakech-Safi region.

Participants will be divided into two groups: an intervention group and a control group. Only the intervention group will receive in-depth training on end-stage renal disease (ESRD), available treatments, potential complications, as well as dietary recommendations and self-care practices tailored for managing arteriovenous fistulas (AVF). The study will assess changes in patients' knowledge, their self-care practices, as well as specific measures such as dry weight, interdialytic weight, and biological markers (calcium, phosphate, and PTH levels).

DETAILED DESCRIPTION:
This study is a randomized controlled trial aimed at evaluating the impact of an educational intervention on improving knowledge, self-care practices, and treatment adherence among hemodialysis patients at the Youssoufia Hemodialysis Center, located in the Marrakech-Safi region.

Methodology: Participants will be recruited from adult patients on hemodialysis for more than three months. They will be randomized into two groups: an intervention group, which will receive educational training, and a control group, which will receive usual care without educational intervention. Sociodemographic and clinical criteria will be collected through the examination of patient medical records.

Intervention: The educational program will consist of six sessions led by a pedagogy expert, in collaboration with a nephrologist a dietitian and hemodialysis nurses. The sessions will cover topics such as end-stage renal disease (ESRD), available treatments, potential complications, as well as dietary recommendations and self-care practices for managing arteriovenous fistulas (AVF).

Evaluations: Outcomes will be measured using validated questionnaires to assess knowledge, self-care practices, and treatment adherence. Biological measures (calcium, phosphate, and PTH levels, dry weight and interdialytic weight) will be taken before the intervention and two months after, in accordance with the center's usual assessments.

The questionnaires will be administered before the intervention and one month after the training to measure changes in patients' knowledge and practices.

Ethical Considerations: The study will adhere to all ethical considerations, including obtaining informed consent and the right for participants to withdraw at any time. The program has already received approval from the ethics committee, and it will also be approved by a nephrologist and a dietitian prior to implementation.

Data Analysis: Data will be analyzed using SPSS. Paired t-tests and independent t-tests will be used to compare results between groups. For non-normally distributed variables, non-parametric tests will be applied. Additionally, linear regression analysis will be conducted to examine associations between variables.

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing hemodialysis (HD) for at least 3 months
* Patients aged > 18 years
* Patients can understand Arabic
* Patients expressing written informed consent to participate in the study

Exclusion criteria :

* Patients with impaired consciousness or memory
* Patients with communication impairments (auditory or verbal)
* Patients with psychological impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Hemodialysis Adherence | Assessed in both groups before the intervention and after one month of intervention.
  * Assessment Tool: End-Stage Renal Disease Adherence Questionnaire (ESRDAQ)
  * Score Range: 0-600
  * Unit: Numerical scale
  * Interpretation: Higher scores indicate better adherence to hemodialysis sessions.
Interdialytic Weight (IDW) | Assessed before the intervention and 2 months after the intervention.
  Assessment Tool: Patients' records Unit: Kilograms (Kg) Measurement Method: Equal to the average of three successive interdialytic weights recorded
Assessment of Patient Knowledge | Assessment before the intervention and after one month, in both groups
  This measure assesses patients' level of knowledge before and after the intervention. the tool used is the litératie questionnaire (specific to hemodialysis patients) by Shih et al. Score ranges from 0 to 26. a high score indicates high knowledge.
Self-Care of the Arteriovenous Fistula | Assessment before the intervention and after 1 months in both groups.
  This measure will examine patients' self-care practices regarding their arteriovenous fistula (AVF) before and after the intervention. The tool is the "scale assessment of self-care behaviors with arteriovenous fistula in hemodialysis" (ASBHD-AVF), with scores ranging from 16 to 80. A high score indicates high-level fistula self-care.
Medication Adherence | Assessed in both groups before the intervention and after one month of intervention.
  * Assessment Tool: End-Stage Renal Disease Adherence Questionnaire (ESRDAQ)
  * Score Range: 0-200
  * Unit: Numerical scale
  * Interpretation: Higher scores indicate better adherence to prescribed medications.
Diet Adherence | Assessed in both groups before the intervention and after one month of intervention.
  * Assessment Tool: End-Stage Renal Disease Adherence Questionnaire (ESRDAQ)
  * Score Range: 0-200
  * Unit: Numerical scale
  * Interpretation: Higher scores indicate better adherence to dietary recommendations
Fluid Restriction Adherence | Assessed in both groups before the intervention and after one month of intervention.
  * Assessment Tool: End-Stage Renal Disease Adherence Questionnaire (ESRDAQ)
  * Score Range: 0-200
  * Unit: Numerical scale
  * Interpretation: Higher scores indicate better adherence to water intake restrictions.
Overall Therapeutic Adherence | Assessed in both groups before the intervention and after one month of intervention
  * Assessment Tool: End-Stage Renal Disease Adherence Questionnaire (ESRDAQ).
  * Score Range: 0-1200
  * Unit: Numerical scale
  * Interpretation: Higher overall scores indicate stronger adherence across all areas.
Dry Weight | Assessed before the intervention (last dry weight) and 2 months after the intervention.
  * Assessment Tool: Patients' records
  * Unit: Kilograms (Kg)
Body Mass Index (BMI) | Calculated before the intervention (using last dry weight) and 2 months after the intervention.
  * Assessment Tool: Derived from patients' records
  * Unit: Kilograms per square meter (Kg/m²)
  * Calculation Method: BMI = Dry Weight (Kg) / Height (m²) using height from patients' records.
Calcium Level | Assessed before the intervention (from the last routine biological assessment) and 2 months after the intervention (from the routine biological assessment taken at least 2 months after the intervention).
  * Assessment Tool: Routine biological assessments (from patients' records)
  * Unit: Millimoles per liter (mmol/L)
Phosphate Level | Assessed before the intervention (from the last routine biological assessment) and 2 months after the intervention (from the routine biological assessment taken at least 2 months after the intervention).
  * Assessment Tool: Routine biological assessments (from patients' records)
  * Unit: Millimoles per liter (mmol/L)
Parathyroid Hormone (PTH) | Assessed before the intervention (from the last routine biological assessment) and 2 months after the intervention (from the routine biological assessment taken at least 2 months after the intervention).
  * Assessment Tool: Routine biological assessments (from patients' records)
  * Unit: Picograms per milliliter (pg/mL)

SECONDARY OUTCOMES:
Assessment of Disease Acceptance. | Assessment before the intervention, in both groups.
  - Assessment of disease acceptance: just before educational intervention. The score ranges from 8 to 40 points; a score of 8 indicates extremely low acceptance of the disease, and 40 indicates extremely high acceptance.
Assessment of Perception of Social Support | Assenssement just before the educational intervention in both groups
  Assessment of perceived social support: just before the intervention, using the Multidimensional Scale of Perceived Social Support, scores range from 12 to 84. Higher scores express stronger feelings of being socially supported

CONTACTS AND LOCATIONS:
Overall Officials: Loubna MAZZI, phD Candidate, Principal Investigator — Laboratory of Pharmacology, Neurobiology, Anthropobiology and Environment, Faculty of Sciences Semlalia, Cadi Ayyad University; Mohamed CHERKAOUI, phD, Study Chair — Laboratory of Pharmacology, Neurobiology, Anthropobiology and Environment, Faculty of Sciences Semlalia, Cadi Ayyad University; Abdelhafid BENKSIM, phd, Study Director — Laboratory of Pharmacology, Neurobiology, Anthropobiology and Environment, Faculty of Sciences Semlalia, Cadi Ayyad University
Locations (1):
- Youssoufia Hemodialysis Center, Youssoufia, Marrakech-Safi Region, Morocco, Youssoufia, Marrakech-Safi, Morocco

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared for several reasons. First and foremost, protecting the confidentiality of participants is a priority. Given the sensitive nature of the data collected, it is essential to ensure that the identity and personal information of participants remain protected.
  Secondly, the logistical requirements associated with preparing the data for sharing can be complex and may require resources that we are unable to mobilize at this time. Finally, we aim to maintain the integrity of the data by limiting access to researchers with the necessary expertise and qualifications to analyze it.
  We are committed to adhering to ethical and regulatory standards for data protection throughout the study.